CLINICAL TRIAL: NCT07041671
Title: Evaluation of Number of Particles Containing Viral RNA and Their Virus Infectivity in Exhaled Air From Participants With Upper Respiratory Tract Infection Symptoms, Before and After Use of One Dose With ColdZyme Mouth Spray
Brief Title: Evaluation Viral RNA and Virus Infectivity in Exhaled Air Before and After Use of One Dose With ColdZyme Mouth Spray
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Enzymatica AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CIV-24-11-049836
Record Dates: First submitted 2025-05-26; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: URTI - Viral Upper Respiratory Tract Infection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ColdZyme treatment (Active Comparator): The subject will use ColdZyme mouth spray once. This will be performed after the first aerosol measurements and before the second.
  Interventions: Device: ColdZyme
- No intervention (No Intervention): Subjects will only perform aerosol measurements, without ColdZyme mouth spray.

INTERVENTIONS:
Device: ColdZyme — ColdZyme is a medical device classified as a Class III device, certified according to the European Medical Devices Regulation (2017/745/EU) (MDR). It has been CE-marked since 2013.
  ColdZyme is a mouth spray that protects against upper respiratory tract viruses causing common cold and flu-like symptoms. ColdZyme forms a protective moisturizing barrier on the mucous membrane of the oral cavity and throat. The viscous barrier catches the virus and thereby the contact between the virus and the epithelial cells are reduced and avoided, thus the barrier disables the viruses' ability to spread and multiply.
  Arms: ColdZyme treatment

SUMMARY:
Many respiratory diseases spread through aerosols. ColdZyme is a mouth spray that protects against upper respiratory tract viruses causing common cold and flu-like symptoms. ColdZyme forms a protective moisturizing barrier on the mucous membrane of the oral cavity and throat. The objective of this study is assessing if ColdZyme could also contribute to decreased airborne transmission by decreasing the amount of (infectious) virus that is exhaled by an infected subject.

DETAILED DESCRIPTION:
The clinical investigation aims to increase the knowledge about the airborne spread of viruses causing upper respiratory tract infections. In particular, it will investigate whether participants with symptoms of a respiratory infection exhale less viruses causing upper respiratory tract infections after using the ColdZyme mouth spray and if the infectivity of exhaled virus particle is reduced. Data from this clinical investigation can possibly show that ColdZyme mouth spray can help reduce the risk of spreading upper respiratory tract virus to the environment.

This is a single centre open label randomized controlled trial. It is an interventional study where subjects are randomized to treatment group (ColdZyme mouth spray) or control group (no spray). The comparison is made between using a mouth spray and not, which cannot be blinded. There are two primary reasons for single centre. Firstly, this is the first study of treatment effects on exhaled viruses and thus feasibility and sensitivity of the methodology is uncertain. Secondly, only a few laboratories internationally have developed instrumentation to perform the measurements.

Subjects enrolled in the study will participate in two different visits, where only visit 1 is related to this clinical investigation regarding ColdZyme. Visit 2 is only for follow-up and the data collected during this visit is not used for investigation of the primary or secondary endpoints, but for explorative analysis that is not related to the hypothesis for ColdZyme. The reason for the second visit is to compare exhaled aerosol characteristics between healthy subjects and subjects with URTI symptoms.

The first visit takes place when the research subject has symptoms of respiratory illness. During the first visit, exhaled aerosol will be collected pre- and post-treatment for the treatment group, and before and after a waiting time of around 20 minutes for the control group. Lung function tests, nasal swabs and questionnaires will be conducted only once per visit and pre-treatment during the first visit.

The exhaled aerosols will be collected into an aerosol sampler (BioSpot, Aerosol Devices Inc.) and analyzed for virus content via qPCR at a later stage. Virus positive samples will be cultured if possible. The particle size distribution and the concentration of exhaled aerosols will be measured directly at the visit by an optical aerosol instrument (OPC, Grimm Aerosol Technik, GmbH). Basic lung function will be measured during both visits by spirometry, oscillometry and AiDA. Symptom scores are collected during both visits.

All measurements are estimated to be made within 2 hours. During the first visit, when the participants have symptoms of respiratory infection, a second sampling of exhaled aerosol will be initiated 20 minutes after use of the mouth spray, or after a waiting time for the control group. The aerosol sampling takes about 30 minutes.

For assessment of the primary variable for the clinical investigation, i.e. virus presence and concentration in the aerosol samples, polymerase chain reaction (PCR) will be used. Maintenance and calibration of the PCR instrument will be performed routinely at the laboratory, for instance by quality control of PCR data from known standard concentrations. Blank aerosol samples will be collected regularly to ensure that there is no cross-contamination or environmental contamination.

The secondary variable, infectivity of virus in the aerosol samples, will be assessed by infecting cell cultures. Negative control wells with uninfected cells will be present in each cell culture plate to ensure that cells were unaffected by other factors.

ELIGIBILITY:
Inclusion criteria for subject selection:

* Male and female subjects above age 18 (inclusive).
* Presence of self-reported sudden onset of at least one of the following symptoms of upper respiratory tract infection case definitions for ILI and ARI (as defined by ECDC (EU 2008, 2012, 2022): Cough, sore throat, shortness of breath, non-allergic rhinitis, fever or feverishness, malaise, headache, myalgia.
* Otherwise of general good health, according to Investigator's judgement.
* Willing and able to give written informed consent for participation in the investigation.

Exclusion criteria for subject selection.

* Known allergy or hypersensitivity to the components of ColdZyme.
* Current use of immunosuppressive therapy within the last 4 weeks prior to Visit 1 and during the investigation.
* Diagnosed chronic respiratory disease that could potentially impact the investigation results, according to Investigator's judgement.
* Self-reported unhealed wounds/mucosal lesions in the mouth and/or throat.
* Participation in another clinical study or investigation within 30 days prior to Visit 1.
* Active smokers
* The Investigator considers the subject unlikely to comply with investigational procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Number of virus genome copies in exhaled aerosol | 20-60 minutes after inhalation of 1 dose treatment of ColdZyme
  Reduction compared to baseline of virus RNA concentrations in exhaled aerosol particles after 1 dose treatment of ColdZyme in subjects in early phase and/or with early common cold/flu-like symptoms (Baseline = virus RNA concentrations in exhaled aerosol particles in untreated participant, i.e before using ColdZyme). RNA copy number is determined by qPCR.

SECONDARY OUTCOMES:
Infectivity of exhaled virus as quantified by TCID50 and MPN | 20-60 minutes after inhalation of 1 dose treatment of ColdZyme
  Infectivity decrease of exhaled virus after 1 dose treatment of ColdZyme in subjects in early phase and/or with early common cold/flu-like symptoms, where the effect is measured in number of infectious virus. Infectivity is quantified by tissue culture infectious dose (TCID50) for screening of infectivity and most probable number MPN for more precise quantification.

CONTACTS AND LOCATIONS:
Locations (1):
- Lund University, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Some individual data will be presented in a table, such as age and gender. Individual data will be shared in a way that individuals can't be identified.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Anonymized IPD and supporting information will be shared upon reasonable request after publication of major findings until at least 10 years after.
Access Criteria: Contact principal investigator Jakob Löndahl (jakob.londahl@design.lth.se) or assoc. prof Malin Alsved (malin.alsved@design.lth.se) for IPD.

REFERENCES:
- [Background] Davison G, Schoeman M, Chidley C, Dulson DK, Schweighofer P, Witting C, Posch W, Matta GG, Consoli C, Farley K, McCullough C, Wilflingseder D. ColdZyme(R) reduces viral load and upper respiratory tract infection duration and protects airway epithelia from infection with human rhinoviruses. J Physiol. 2025 Mar;603(6):1483-1501. doi: 10.1113/JP288136. Epub 2025 Feb 28. PMID 40019230